CLINICAL TRIAL: NCT04371744
Title: QT-Logs : a Clinical Study to Monitor Cardiac Safety, With Artificial Intelligence for QT Interval Analysis of ECG Data From Smartwatches, in Patients Receiving Hydroxychloroquine Treatment for COVID-19
Brief Title: QT-Logs : Artificial Intelligence for QT Interval Analysis of ECG From Smartwatches in Patient Receiving Treatment for Covid-19
Acronym: QT-Logs
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: CIL 2020-52
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational pilot prospective study will evaluate a new method for remote monitoring of corrected QT measurement using an artificial intelligence (AI)-based solution and ECG data collected via smartwatches (AI-QTc), in patients ambulatory treated with the HC-AZ combination, at the early stage of COVID-19 infection, at a tertiary hospital center. Daily ECGs will be performed via the smartwatches. AI-QTc will be compared to standard manual QTc reviewed by cardiologist. Correlation and agreement between measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* SARS-COV-2 confirmed infection by positive nasopharyngual PCR
* Prescription of association hydroxychloroquine and azythromycine for COVI-19 therapy
* Patient's smartphone able to download the smartwatches application

Exclusion Criteria:

* Presence of a pacemaker
* Pregnant or breastfeeding females
* Refusal to participate
* Incapacity
* Adult under legal protection (trusteeship, guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutives patients ambulatory treated with the Hydroxychloroquine and Azythromycine combination, at the early stage of COVID-19 infection for 10 days, at the university hospital of La Timone, in Marseille
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Corrected QT (QTc) interval measurement | 10 days
  Measurement of QTc using an artificial intelligence (AI)-based solution and ECG data collected via smartwatches, compare to standard 12 leads ECG reviewed by cardiologist

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Maille B, Wilkin M, Million M, Resseguier N, Franceschi F, Koutbi-Franceschi L, Hourdain J, Martinez E, Zabern M, Gardella C, Tissot-Dupont H, Singh JP, Deharo JC, Fiorina L. Smartwatch Electrocardiogram and Artificial Intelligence for Assessing Cardiac-Rhythm Safety of Drug Therapy in the COVID-19 Pandemic. The QT-logs study. Int J Cardiol. 2021 May 15;331:333-339. doi: 10.1016/j.ijcard.2021.01.002. Epub 2021 Jan 29. PMID 33524462